CLINICAL TRIAL: NCT00256893
Title: A Randomised, Double Blind, Placebo-controlled, Parallel Group Study to Investigate the Safety and Efficacy of Controlled-release Ropinirole (CR) (1-24 mg) Administered Once Daily for 12 Weeks in Subjects With Fibromyalgia
Brief Title: Fibromyalgia Study In Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROF102100
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Fibromyalgia Syndrome, Primary
Keywords: pain intensity; numerical rating scale; fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — ropinirole

INTERVENTIONS:
Drug: ropinirole

SUMMARY:
A study to investigate ropinirole for treatment of the symptoms of fibromyalgia and in particular the widespread pain associated with this condition. A total 160 subjects (80 per treatment arm) are being recruited from approximately 25 centres in 9 European countries. Male and female subjects greater than 18 years of age with a diagnosis of primary fibromyalgia, as defined by the American College of Rheumatology (ACR) criteria, are eligible for study entry. Subjects will receive either ropinirole (1-24mg) or placebo, depending upon a statistically defined allocation to treatment. The primary endpoint is improvement in pain score by 12 weeks of treatment. An 11 point numerical rating scale for the assessment of the subject's pain is being collected on a daily diary. In addition, the overall improvement in quality of life for the subject will be assessed by means of a number of subject-completed questionnaires during the treatment period. Safety of the treatment regimen will be assessed throughout the study.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of primary fibromyalgia as defined by the American College of Rheumatology (ACR).
* Females of childbearing potential will only be eligible if taking adequate contraceptive measures.
* Other co-existent chronic pain conditions such as osteoarthritis, will not exclude the subject if the pain associated with the condition is less severe than the pain of fibromyalgia.
* Only subjects experiencing moderate/severe pain (pain intensity score >= 4 on the pain numerical rating scale) will be eligible for this study.
* Subjects that are generally well.
* Have the ability to discontinue prohibited medications for the duration of the study.

Exclusion criteria:

* Subjects with 'flare' of arthritic conditions.
* Evidence of clinically significant medical conditions including cardiovascular conditions (e.g. postural hypotension, and raised blood pressure, ECG abnormalities).
* History of drug and/or alcohol abuse or major depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164
Dates: Start 2004-11; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity score from baseline to last week of treatment (week 12)

SECONDARY OUTCOMES:
Pain relief. Global function: PGIC (Patient Global Impression of Change)and CGIC (Clinical Global Impression of Change), FIQ (Fibromyalgia Impact Questionnaire), Pain severity and impact on physical function, Sleep quality, tender pointpressure threshold

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Diepenbeek
  - GSK Investigational Site, Merksem
- GSK Investigational Site, Frederiksberg, Denmark
- Finland (3):
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Mikkeli
- France (2):
  - GSK Investigational Site, Lomme
  - GSK Investigational Site, Paris
- Germany (4):
  - GSK Investigational Site, Fellbach, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Bad Hersfeld, Hesse
  - GSK Investigational Site, Hüttenberg, Hesse
- Italy (3):
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
- GSK Investigational Site, Zwolle, Netherlands
- GSK Investigational Site, Mölndal, Sweden
- United Kingdom (3):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Truro, Cornwall
  - GSK Investigational Site, Poole, Dorset

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: ROF102100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ROF102100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ROF102100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ROF102100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ROF102100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ROF102100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ROF102100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register